CLINICAL TRIAL: NCT02420327
Title: The Use of Low-Dose Galantamine to Potentiate the Attention-Enhancing Effects of Low-Dose Nicotine
Brief Title: Low-Dose Galantamine to Potentiate the Attention-Enhancing Effects of Low-Dose Nicotine
Acronym: GalaNic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Britta Hahn, Associate Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Basic Science
Other Study IDs: HP-00057097
Record Dates: First submitted 2015-04-14; First posted 2015-04-17 (Estimated); Results first posted 2018-08-17 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Basic Science Study of the Mechanisms of Attentional Enhancement by Compounds Acting on the Nicotinic Receptor
Keywords: nicotine; galantamine; attention; cognition; non-smoker
MeSH Terms: interventions — Galantamine; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo patch and placebo capsule (Experimental): On the double-placebo test day, participants receive a placebo patch and a placebo capsule.
  Interventions: Drug: Placebo patch & placebo capsule
- Nicotine patch and placebo capsule (Experimental): On the nicotine test day, participants receive a nicotine patch (7 mg/24 hrs) and a placebo capsule.
  Interventions: Drug: Nicotine patch & placebo capsule
- Placebo patch and galantamine capsule (Experimental): On the galantamine test day, participants receive a placebo patch and a capsule containing 4 mg of galantamine.
  Interventions: Drug: Placebo patch & galantamine capsule
- Nicotine patch and galantamine capsule (Experimental): On the nicotine + galantamine test day, participants receive a nicotine patch (7 mg/24 hrs) and a capsule containing 4 mg of galantamine.
  Interventions: Drug: Nicotine patch and galantamine capsule

INTERVENTIONS:
Drug: Placebo patch & placebo capsule — On this test day, cognition is assessed after administration of a placebo patch and a placebo capsule.
  Arms: Placebo patch and placebo capsule
Drug: Placebo patch & galantamine capsule — On this test day, cognition is assessed after administration of a placebo patch and a galantamine capsule (4 mg p.o.).
  Arms: Placebo patch and galantamine capsule
Drug: Nicotine patch & placebo capsule — On this test day, cognition is assessed after administration of a nicotine patch (7 mg/24 hrs) and a placebo capsule.
  Arms: Nicotine patch and placebo capsule
Drug: Nicotine patch and galantamine capsule — On this test day, cognition is assessed after administration of a nicotine patch (7 mg/24 hrs) and a galantamine capsule (4 mg p.o.).
  Arms: Nicotine patch and galantamine capsule

SUMMARY:
The aim of this study is to test whether the attention-enhancing effects of low-dose nicotine can be enhanced by the drug galantamine, FDA-approved for the treatment of Alzheimer's disease. This proof-of-principle study is performed in healthy non-smokers and involves two single exposures to a nicotine patch (7 mg/24 hrs) and two single exposures to galantamine (4 mg). The dose of galantamine is substantially lower than the clinical dose range of 16-24 mg/day. The hypothesis is that performance-enhancing effects of nicotine are greater in the presence of this low dose of galantamine.

DETAILED DESCRIPTION:
Healthy non-smokers will be screened for study eligibility and receive training on three different attention tasks. Over four test session, participants will then perform these tasks after receiving (1) a placebo patch and a placebo capsule, (2) a nicotine patch (7 mg/24 hrs) and a placebo capsule, (3) a placebo patch and a galantamine capsule, and (4) a nicotine patch and a galantamine capsule. The four test session are performed on separate days and take approximately 7 hours each. During the first 5 hours, the participant may read or watch TV while nicotine and/or galantamine are being absorbed. During the last two hours, the participant will perform the attention tasks on a computer. The investigators hypothesize that performance-enhancing effects of nicotine, which were documented in previous research, will be larger in the presence than in the absence of galantamine. This proof-of-concept would have implications for the development of drugs for the treatment of conditions such as Alzheimer's disease or schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* Aged 21 to 55 years.
* No exposure to any nicotine-containing product in the last year.
* Smoked no more that 40 cigarettes, cigars or cigarillos in lifetime.
* Normal or corrected to normal vision (at least 20/80).
* Body weight 110-220 lbs.

Exclusion Criteria:

* Pregnant or breast-feeding.
* Drug or alcohol abuse or dependence currently or in the last 2 years.
* DSM Axis I mood, anxiety or psychotic disorder.
* Cardiovascular or cerebrovascular disease, such as history of myocardial infarction and ischemia, heart failure, angina, stroke, severe arrhythmias, or EKG abnormalities (Wolf-Parkinson-White syndrome, Complete left bundle branch block, PR interval <120 ms or >200 ms, Prolonged QT interval (corrected) >500 ms, Cardiac arrhythmias as defined by PACs >3 per min or PVCs >1 per min).
* Uncontrolled hypertension (resting systolic BP above 140 or diastolic above 90 mm Hg).
* Hypotension (resting systolic BP below 90 or diastolic below 60).
* Significant kidney or liver impairment.
* Moderate to severe asthma.
* Obstructive pulmonary disease.
* Type I or II diabetes.
* Use of any centrally active medications; any peripherally acting cholinergic medications; cimetidine; ketoconazole; erythromycin; quinidine, or chronic nonsteroidal anti-inflammatory drugs.
* History of or current neurological illnesses, such as stroke, seizure disorders, neurodegenerative diseases, or organic brain syndrome.
* Learning disability, mental retardation, or any other condition that impedes cognition.
* Heart rate <55 bpm.
* Current or history of gastric ulcer disease.
* Any surgeries requiring full anesthesia scheduled within 2 weeks of any of the study test sessions.
* Anemia.
* Inability to perform the Rapid Visual Information Processing Task.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-09; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Britta Hahn, Ph.D., Principal Investigator — University of Maryland, Baltimore
Locations (1):
- University of Maryland School of Medicine, Maryland Psychiatric Research Center, Catonsville, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Adults: All participants receive the following four interventions, on separate days, in a counterbalanced order:
  1. placebo patch and placebo capsule
  2. placebo patch and galantamine capsule
  3. nicotine patch and placebo capsule
  4. nicotine patch and galantamine capsule
  Placebo patch & placebo capsule: On this test day, cognition is assessed after administration of a placebo patch and a placebo capsule.
  Placebo patch & galantamine capsule: On this test day, cognition is assessed after administration of a placebo patch and a galantamine capsule (4 mg p.o.).
  Nicotine patch & placebo capsule: On this test day, cognition is assessed after administration of a nicotine patch (7 mg/24 hrs) and a placebo capsule.
  Nicotine patch and galantamine capsule: On this test day, cognition is assessed after administration of a nicotine patch (7 mg/24 hrs) and a galantamine capsule (4 mg p.o.).
Period: Overall Study
Arm/Group | Healthy Adults
Started | 43
Completed | 27
Not Completed | 16
Not completed — Adverse Event | 7
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 1
Not completed — Protocol Violation | 1

BASELINE CHARACTERISTICS:
Population: This includes 27 study completers and 16 study non-completers.
Arm/Group | Healthy Adults
Number analyzed (Participants) | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 38
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 18
  White | 18
  More than one race | 3
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Spatial Attentional Resource Allocation Task Predictive Trials Reaction Time
Description: The task requires detecting brief target stimuli presented at one of four locations in the four corner of the screen. On predictive trials, a central cue predicts the target location.
Time Frame: 45 min
Population: 27 healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 27 | 27 | 27 | 27
ms | 420 (66) | 408 (56) | 416 (61) | 413 (63)

2. Primary Outcome: Rapid Visual Information Processing Task Hit Rate
Description: The task requires following a stream of digits and detecting three consecutive odd or even numbers. The Hit Rate reflects the percentage of all target sequences that were detected.
Time Frame: 30 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: percentage of all targets
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 27 | 27 | 27 | 27
percentage of all targets | 50 (19) | 54 (18) | 49 (21) | 54 (19)

3. Primary Outcome: Change Detection Task Accuracy
Description: The task requires encoding the color of 1 or 5 shape items and reporting whether or not one of the items changed color. Accuracy refers to the percentage of all trials in which a correct response was given.
  One participant's data were excluded from this task because of excessive no-response trials.
Time Frame: 15 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: percentage of all trials
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 26 | 26 | 26 | 26
percentage of all trials | 83 (6) | 83 (6) | 84 (6) | 84 (6)

4. Primary Outcome: Spatial Attentional Resource Allocation Task (SARAT) Non-predictive Trial Reaction Time
Description: The task requires responding to brief target stimuli presented randomly in one of four locations in the four corners of the screen. On non-predictive trial, the cue does not provide any advance information about where the target will occur.
Time Frame: 45 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 27 | 27 | 27 | 27
ms | 472 (71) | 455 (62) | 465 (66) | 449 (64)

5. Primary Outcome: Rapid Visual Information Processing Task Reaction Time
Description: The task requires the detection of three consecutive odd or three consecutive even digits in a stream of sequentially presented digits.
Time Frame: 30 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 27 | 27 | 27 | 27
ms | 463 (59) | 459 (64) | 473 (70) | 459 (63)

6. Primary Outcome: Change Detection Task Reaction Time
Description: The task requires encoding the color of 1 or 5 shape items and reporting whether or not one of the items changed color.
  One participant's data were excluded from this task because of excessive no-response trials.
Time Frame: 15 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 26 | 26 | 26 | 26
ms | 1018 (241) | 1023 (216) | 1043 (239) | 973 (225)

7. Secondary Outcome: Profile of Mood Scale - Total Mood Disturbance
Description: Participants rate their current subjective state on a list of adjectives, which contribute to six factors/subscales. "Total Mood Disturbance" is a composite measure, obtained by summing the scores of all subscales, each with a range of 0-4, weighting the one positively valenced factor negatively. Thus, smaller or more negative values represent a more positive mood state. The theoretical range of the "Total Mood Disturbance" measure is from -4 to +20.
Time Frame: 5 min
Population: Healthy adult non-smokers
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
Number analyzed (Participants) | 27 | 27 | 27 | 27
score on a scale | -0.32 (0.91) | -0.48 (0.98) | -0.60 (0.99) | -0.43 (1.16)

ADVERSE EVENTS:
Time Frame: During each of the four test sessions (7 hours each).
Description: Participants had vital signs taken and completed a side-effects checklist hourly (after patch) or every thirty minutes (after capsule). Unsolicited reports of adverse effects were also recorded.
Arm/Group | Placebo Patch and Placebo Capsule | Nicotine Patch and Placebo Capsule | Placebo Patch and Galantamine Capsule | Nicotine Patch and Galantamine Capsule
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34 | 0/30 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34 | 0/30 | 0/32
Other Adverse Events (participants affected / at risk) | 1/32 | 5/34 | 0/30 | 4/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Patch and Placebo Capsule (N=32) | Nicotine Patch and Placebo Capsule (N=34) | Placebo Patch and Galantamine Capsule (N=30) | Nicotine Patch and Galantamine Capsule (N=32)
vomiting (Gastrointestinal disorders) | 0 (0) | 4 (4) | 0 (0) | 4 (4)
nausea (Gastrointestinal disorders) | 0 (0) | 5 (5) | 0 (0) | 4 (4)
palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
pain at patch site (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-03): https://cdn.clinicaltrials.gov/large-docs/27/NCT02420327/Prot_SAP_000.pdf